CLINICAL TRIAL: NCT00606463
Title: Gen2 Cardiac Ablation System Isthmus-Dependent Atrial Flutter Study
Brief Title: Gen2 Isthmus-Dependent Atrial Flutter Ablation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Abbott funding allocated to a different project.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0611.1
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- (Gen2 Cardiac Ablation System) (Experimental): Ablation of isthmus-dependent atrial flutter
  Interventions: Device: Cardiac Ablation (Gen2 Cardiac Ablation System)

INTERVENTIONS:
Device: Cardiac Ablation (Gen2 Cardiac Ablation System) — Ablation of isthmus-dependent atrial flutter

SUMMARY:
Irrigated catheter for ablation of isthmus-dependent atrial flutter

DETAILED DESCRIPTION:
This study intends to use an investigational irrigated catheter for ablation of isthmus-dependent atrial flutter

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ablation of isthmus-dependent atrial flutter

Exclusion Criteria:

* Prior ablation of isthmus-dependent atrial flutter
* Atypical or scar flutter
* Significant heart disease
* Intracardiac thrombus
* Prior cardiac surgery (within 1 month)
* Contraindication to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incidence of intraprocedural, serious cardiac adverse event | 7 days post-procedure
  Defined as the Incidence of intraprocedural, serious cardiac adverse event

OTHER OUTCOMES:
Bi-direction block and non-inducibility of atrial flutter | Procedural
  Acute Procedure success defined as bi-directional block and non-inducibility of atrial flutter

CONTACTS AND LOCATIONS:
Overall Officials: Vance Plumb, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama Birmingham, Birmingham, Alabama
  - St. Barnabus Medical Center, West Orange, New Jersey
  - Doylestown Hospital, Doylestown, Pennsylvania

IPD SHARING:
Plan to Share IPD: No